CLINICAL TRIAL: NCT01267227
Title: Effect of Pterostilbene on Cholesterol, Blood Pressure and Oxidative Stress
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Mississippi Medical Center (Other)
Responsible Party: Principal Investigator, Daniel Riche, Assistant Professor of Pharmacy Practice and Medicine, University of Mississippi Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2010-0225
Record Dates: First submitted 2010-12-17; First posted 2010-12-28 (Estimated); Results first posted 2013-05-03 (Estimated); Last update posted 2018-01-10 (Actual); Status verified 2017-12

CONDITIONS: Hyperlipidemia; Blood Pressure; Oxidative Stress
Keywords: Hyperlipidemia; Cholesterol; Blood Pressure; Oxidative Stress; Pterostilbene; Blueberry; Grape Extract
MeSH Terms: conditions — Hyperlipidemias | interventions — Pterocarpus marsupium; whole grape extract

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- High Dose (Active Comparator): Pterostilbene 125 mg twice daily
  Interventions: Drug: Pterostilbene 125 mg twice daily
- Low Dose (Active Comparator): Pterostilbene 50 mg twice daily
  Interventions: Drug: Pterostilbene 50 mg twice daily
- Low Dose Combination (Active Comparator): Pterostilbene 50 mg/Grape Extract 100 mg twice daily
  Interventions: Drug: Pterostilbene 50 mg twice daily; Drug: Grape Extract
- Placebo (Placebo Comparator): Matching placebo twice daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pterostilbene 50 mg twice daily — Pterostilbene 50 mg twice by mouth daily for 6 to 8 weeks
  Other Names: pTeroPure
  Arms: Low Dose; Low Dose Combination
Drug: Placebo — Matching placebo by mouth twice daily for 6 to 8 weeks
  Arms: Placebo
Drug: Grape Extract — Grape extract 100 mg twice daily for 6-8 weeks
  Other Names: ShanStar Concord Grape
  Arms: Low Dose Combination
Drug: Pterostilbene 125 mg twice daily — Pterostilbene 125 mg twice daily for 6-8 weeks
  Other Names: pTeropure
  Arms: High Dose

SUMMARY:
Pterostilbene is one of several stilbenes found in certain berries, particularly blueberries, that have demonstrated pre-clinical benefit to cholesterol, blood pressure, and oxidative stress. The purpose of this study is to evaluate whether pterostilbene will help control cholesterol and blood pressure, as well as improve markers for oxidative stress in patients with dyslipidemia meeting inclusion criteria. The investigators also want to look at the safety of pterostilbene in these patients.

DETAILED DESCRIPTION:
Subjects will be divided into one of four groups: (1) pterostilbene 50 mg twice daily; (2) pterostilbene 125 mg twice daily; (3) pterostilbene 50 mg/grape extract 100 mg twice daily; (4) matching placebo twice daily taken either one hour before or two hours after a meal. Blood and urine will be collected at enrollment and final study visits. If the patient's low density lipoprotein-C (LDL-C) or total cholesterol (TC) is not within the inclusion criteria based on enrollment blood drawn, the patient will not be allowed to initiate study medication. All study visits will consist of brief clinical examination (including vital signs), subjective adverse event reporting, and fasting donated blood and urine for clinical laboratory tests. Pill counts will be done to assess compliance.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥18 years of age with a previous TC ≥200 mg/dL and/or a LDL ≥100 mg/dL on either no therapy or stable therapy
* Any concomitant cholesterol medication (not listed in the exclusion criteria) must be at a stable dose for at least 2 months prior to baseline laboratory

Exclusion Criteria:

* Patients with significant hepatic, renal or gastrointestinal tract disease
* Receiving thiazolidinediones or fibric acid derivatives
* Current overt cardiovascular disease
* Women of reproductive potential not receiving birth control
* Pregnant/nursing women

Ages: 18 Years to 88 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2010-12; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel M Riche, Pharm.D., Principal Investigator — University of Mississsippi
Locations (1):
- University of Mississippi Medical Center, Jackson, Mississippi, United States

REFERENCES:
- [Background] Paul S, Rimando AM, Lee HJ, Ji Y, Reddy BS, Suh N. Anti-inflammatory action of pterostilbene is mediated through the p38 mitogen-activated protein kinase pathway in colon cancer cells. Cancer Prev Res (Phila). 2009 Jul;2(7):650-7. doi: 10.1158/1940-6207.CAPR-08-0224. Epub 2009 Jun 23. PMID 19549798
- [Background] Rimando AM, Kalt W, Magee JB, Dewey J, Ballington JR. Resveratrol, pterostilbene, and piceatannol in vaccinium berries. J Agric Food Chem. 2004 Jul 28;52(15):4713-9. doi: 10.1021/jf040095e. PMID 15264904
- [Background] Rimando AM, Nagmani R, Feller DR, Yokoyama W. Pterostilbene, a new agonist for the peroxisome proliferator-activated receptor alpha-isoform, lowers plasma lipoproteins and cholesterol in hypercholesterolemic hamsters. J Agric Food Chem. 2005 May 4;53(9):3403-7. doi: 10.1021/jf0580364. PMID 15853379
- [Background] Amarnath Satheesh M, Pari L. The antioxidant role of pterostilbene in streptozotocin-nicotinamide-induced type 2 diabetes mellitus in Wistar rats. J Pharm Pharmacol. 2006 Nov;58(11):1483-90. doi: 10.1211/jpp.58.11.0009. PMID 17132211
- [Background] Satheesh AM, Pari L. Effect of pterostilbene on lipids and lipid profiles in streptozotocin-nicotinamide induced type 2 diabetes mellitus. Journal of Applied Biomedine 6(1):31-37, 2008.
- [Result] Riche DM, Riche KD, Blackshear CT, McEwen CL, Sherman JJ, Wofford MR, Griswold ME. Pterostilbene on metabolic parameters: a randomized, double-blind, and placebo-controlled trial. Evid Based Complement Alternat Med. 2014;2014:459165. doi: 10.1155/2014/459165. Epub 2014 Jun 25. PMID 25057276
- [Result] Riche DM, McEwen CL, Riche KD, Sherman JJ, Wofford MR, Deschamp D, Griswold M. Analysis of safety from a human clinical trial with pterostilbene. J Toxicol. 2013;2013:463595. doi: 10.1155/2013/463595. Epub 2013 Feb 4. PMID 23431291

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Medical clinic
Period: Overall Study
Arm/Group | High Dose | Low Dose | Low Dose Combination | Placebo
Started | 20 | 20 | 20 | 20
Completed | 19 | 19 | 18 | 17
Not Completed | 1 | 1 | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | High Dose | Low Dose | Low Dose Combination | Placebo | Total
Number analyzed (Participants) | 20 | 20 | 20 | 20 | 80
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 16 | 19 | 17 | 17 | 69
  >=65 years | 4 | 1 | 3 | 3 | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.6 (11.2) | 53.6 (7.9) | 53.0 (13.7) | 54.4 (11.9) | 53.6 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 15 | 15 | 13 | 57
  Male | 6 | 5 | 5 | 7 | 23
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 20 | 20 | 80

OUTCOME MEASURES:

1. Primary Outcome: LDL
Description: Increase in low density lipoprotein (LDL)
Time Frame: Baseline and 6-8 weeks
Measure: Mean (95% Confidence Interval); unit: mg/dL
Groups:
- High Dose: Pterostilbene 125 mg twice daily. Unadjusted change from baseline.
- Low Dose: Pterostilbene 50 mg twice daily. Unadjusted change from baseline.
- Low Dose Combination: Pterostilbene 50 mg/Grape Extract 100 mg twice daily. Unadjusted change from baseline.
- Placebo: Matching placebo twice daily. Unadjusted change from baseline.
Arm/Group | High Dose | Low Dose | Low Dose Combination | Placebo
Number analyzed (Participants) | 20 | 20 | 20 | 20
mg/dL | 19.67 [5.28 to 34.05] | 20.04 [5.68 to 34.40] | 5.33 [-9.16 to 19.82] | 0 [0 to 0]

2. Secondary Outcome: Blood Pressure
Description: Reduction in systolic blood pressure versus placebo
Time Frame: 6-8 weeks
Measure: Mean (95% Confidence Interval); unit: mmHg
Arm/Group | High Dose | Low Dose | Low Dose Combination | Placebo
Number analyzed (Participants) | 20 | 20 | 20 | 20
mmHg | 7.77 [2.38 to 13.17] | 3.67 [-1.74 to 9.09] | 6.72 [1.25 to 12.18] | 0 [0 to 0]

3. Secondary Outcome: Subjective Adverse Effects
Description: Number of participants with adverse effects as a measure of safety
Time Frame: Baseline and 6-8 weeks
Measure: Number; unit: participants
Arm/Group | High Dose | Low Dose | Low Dose Combination | Placebo
Number analyzed (Participants) | 20 | 20 | 20 | 20
participants | 5 | 3 | 2 | 2

ADVERSE EVENTS:
Arm/Group | High Dose | Low Dose | Low Dose Combination | Placebo
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 5/20 | 3/20 | 2/20 | 2/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | High Dose (N=20) | Low Dose (N=20) | Low Dose Combination (N=20) | Placebo (N=20)
GI (Gastrointestinal disorders) | 4 (4) | 1 (1) | 1 (1) | 1 (1)
Muscle Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Itching (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Disclosure of the submitted materials approved per contractual agreement.